CLINICAL TRIAL: NCT04459377
Title: An Analysis of Ketamine Analgesia in Third Molar Surgery -Effects, Safety and Influence on Inflammatory Biomarkers in Plasma
Brief Title: Ketamine Analgesia in Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Uppsala University (Other); Center for Clinical Research Dalarna, Sweden (Other)
Responsible Party: Principal Investigator, Lars Eriksson, Senior Consultant in Oral and Maxillofacial Surgery, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140929sketamine; 2014-004235-39 (EudraCT Number)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pain; Postoperative
Keywords: Ketamine; Postoperative; Pain management; Third molar
MeSH Terms: conditions — Pain; Agnosia | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Sodium Chloride solution (9mg / ml) 0.2ml / kg slow intravenous injection (2ml / min).
  Interventions: Drug: Sodium Chloride 0.9% Inj
- K1 (Active Comparator): S-Ketamine (0.125 mg / kg body weight). (0.625mg / ml x 0.2ml / kg) slow intravenous injection (2ml / min).
  Interventions: Drug: S-Ketamine
- K2 (Active Comparator): S-Ketamine (0.25 mg / kg body weight). (1.25mg / ml x 0.2ml / kg) slow intravenous injection (2ml / min).
  Interventions: Drug: S-Ketamine

INTERVENTIONS:
Drug: S-Ketamine — Patients are randomized to three groups. Randomization in blocks of six patients stratified by sex. A list of serial numbers and randomized group affiliation is produced which is open to the pharmacy's manufacturing staff and closed to the staff of the trial. The pharmacy prepares filled syringes with investigation drug in accordance with randomized group affiliation.
  All groups are sedated with midazolam intravenously to a defined end point. A syringe pump with volume accuracy ± 2% injects the test drug (P, K1 or K2). One infusion set is coupled between the syringe and a three-way connection, which in turn is connected to a peripheral venous catheter (PVK). This PVK is also used for blood sampling. Blood is sampled at two occasions. Directly preoperatively and two hours after surgery. The third molar is surgically removed.
  Arms: K1; K2
Drug: Sodium Chloride 0.9% Inj — Patients are randomized to three groups. Randomization in blocks of six patients stratified by sex. A list of serial numbers and randomized group affiliation is produced which is open to the pharmacy's manufacturing staff and closed to the staff of the trial. The pharmacy prepares filled syringes with investigation drug in accordance with randomized group affiliation.
  All groups are sedated with midazolam intravenously to a defined end point. A syringe pump with volume accuracy ± 2% injects the test drug (P, K1 or K2). One infusion set is coupled between the syringe and a three-way connection, which in turn is connected to a peripheral venous catheter (PVK). This PVK is also used for blood sampling. Blood is sampled at two occasions. Directly preoperatively and two hours after surgery. The third molar is surgically removed.
  Arms: Placebo

SUMMARY:
BACKGROUND AND PURPOSE Outpatient surgery (day case surgery) is increasing. When the patients go home on the same day, this demands safe pain relief. A reduction of morphine (opioid) use is sought because of side effects and the dependency risk. An effective alternative to opioids is ketamine, which lacks the side effects of opioids but provides powerful analgesic effects.

METHOD At the start of surgery, Ketamine or placebo will be given in a vein to evaluate if the acute pain decreases significantly. Inflammation is known to cause pain. By measuring different proteins in the blood, the investigators want to understand how inflammation links to the pain. Wisdom tooth surgery provides significant post-operative pain and is a widely accepted pain model in drug studies. Patients referred for wisdom tooth surgery are asked to participate in the study. For statistical certainty, in total 165 persons will be enrolled to three groups. Two with active drug (different dose) and one placebo. Everyone gets local anesthesia. The completion of the study will be done in four years. The Ethics Review Board has approved the study.

CLINICAL RELEVANCE Effective pain relief after daily surgical procedures is important for patient´s safety and reducing the risk of long-term pain. It is also ethically necessary for the continued expansion of day case surgery. New knowledge of the mechanisms of pain increases the opportunities for individual and safe pain relief. Day case surgery is performed in all operating specialties, this might affects many patients nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or mild well-compensated systemic disease (ASA I & II)
* 18- <45 years
* 50-100 kg body weight

Exclusion Criteria:

* Medication drugs: analgesics, hypnotics (the last week before surgery), thyroid hormones, psychoactive drugs or monoamine oxidase inhibitors (MAO inhibitors).
* Hypertension [> 150/95 mmHg in screening study]
* Heart failure
* Psychosis
* Epilepsy
* Hyperthyreosis
* Myasthenia gravis
* Glaucoma
* Verified sleep apnea
* Diabetes (insulin treated)
* Porphyria
* Pregnancy
* Breast-feeding
* Blood transmitted infections, such as HIV and hepatitis B and C
* Known hypersensitivity to midazolam, ketamine, ibuprofen, or local anesthetics
* Inability to obtain the requisite written or oral information

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | 4 hours postoperatively
  Postoperative pain measured by Visual analog scale (VAS). From minimum 0mm to maximum 100mm. 0mm is no pain and 100mm is worst pain imaginable. Changes in Visual Analog Scale value from preoperatively to 4 hours postoperatively

SECONDARY OUTCOMES:
Safety (Oxygen saturation) | Up to 2 hours.
  Change in oxygen saturation measured by pulseoximeter %. Intra individually and between the groups. From start to completion of the ketamine infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sand, Professor, DDS, MD, Study Director — Uppsala University
Locations (1):
- Käkkirurgiska kliniken, Falu lasarett, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eriksson LB, Larsson A, Eriksson M, Tegelberg A, Thor A, Gordh T. Methodological comparison between salivary and plasma inflammatory biomarkers in third molar surgery patients. BMC Oral Health. 2025 Nov 22;25(1):1902. doi: 10.1186/s12903-025-07368-2. PMID 41272580